CLINICAL TRIAL: NCT02950428
Title: ACURATE Neo™ Aortic Bioprosthesis for Implantation Using the ACURATE Neo™ TA Transapical Delivery System in Patients With Severe Aortic Stenosis
Brief Title: ACURATE Neo™ TA Delivery System in Patient With Severe Aortic Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Symetis SA (Industry)
Responsible Party: Sponsor
Organization: Boston Scientific Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-01
Record Dates: First submitted 2016-02-12; First posted 2016-11-01 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Aortic Stenosis
Keywords: TAVI; Aortic Stenosis; transcatether Aortic Valve Implantation
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACURATE neo™TA Delivery System (Experimental): Patients implanted with ACURATE neo™ Aortic Bioprosthesis and ACURATE neo™ TA Transapical Delivery System
  Interventions: Device: ACURATE neo™TA Delivery System

INTERVENTIONS:
Device: ACURATE neo™TA Delivery System — ACURATE neo™ Aortic Bioprosthesis and ACURATE neo™TA Transapical Delivery System on patients with severe aortic stenosis where conventional aortic valve replacement (AVR) via open-heart surgery is considered to be high risk

SUMMARY:
The purpose of this investigation is to collect data pertaining to the safety and performance of the ACURATE neo (TM) Aortic Bioprosthesis as implanted with the ACURATE neo (TM) TA Transapical Delivery System. This device is intended for treatment of subjects with severe aortic stenosis (AS) who have high risk for conventional aortic valve replacement (AVR) surgery. The ACURATE neo (TM) Aortic Bioprosthesis is intended for use via minimally-invasive transapical implantation in a well-defined population.

DETAILED DESCRIPTION:
This is a single arm, prospective, multicenter non randomised and open trial of the treatment of patients with severe aortic stenosis where conventional aortic valve replacement (AVR) via open heart surgery is considered to be high risk. All patients will be followed up to 5 years after the intervention.

The primary objective is to evaluate the safety and performance of the study device in patients presenting with severe aortic stenosis considered to be high risk for surgery Secondary objective is to evaluate adverse events and study device performance.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years old
2. Severe aortic stenosis defined as:

   * Mean aortic gradient > 40 mmHg or
   * Peak jet velocity > 4.0 m/s or
   * Aortic valve area of < 0.8 cm2
3. High risk patient determined by a multidisciplinary heart team consensus (cardiologist and cardiac surgeon) that patient is not a surgical candidate for conventional AVR due to risk factors such as STS Score (8% or higher) or other co-morbid conditions unrelated to aortic stenosis such as severe chronic obstructive pulmonary disease (COPD), chest deformities and irradiated mediastinum
4. NYHA Functional Class > II
5. Multidisciplinary heart team (cardiologist and cardiac surgeon) consensus that the transapical approach is the most suitable access route for TAVI due to the presence of the following anatomic conditions:

   * porcelain aorta or
   * severely calcified or highly tortuous peripheral vasculature not appropriate for transfemoral transcatheter aortic valve implantation or
   * vessels too small for retrograde approach or
   * other anatomical conditions making transapical approach more suitable
6. Aortic annulus diameter from ≥ 21mm up to ≤ 27mm by CT or TEE
7. Patient willing to participate in the study and provides signed informed consent

Exclusion Criteria:

1. Congenital unicuspid or bicuspid aortic valve or non-calcified
2. Extreme eccentricity of calcification
3. Severe mitral regurgitation (> Grade 3)
4. Pre-existing prosthetic heart valve in any position and / or prosthetic ring
5. LV apex is not accessible via transapical access due to severe chest deformity
6. Previous surgery of the LV using a patch, such as the Dor procedure
7. Presence of apical LV thrombus
8. Calcified pericardium
9. Septal hypertrophy unacceptable for transapical procedure
10. Transesophageal echocardiogram (TEE) is contraindicated
11. ECHO evidence of intracardiac mass, thrombus, or vegetation
12. LVEF < 20% by ECHO
13. Need for emergency intervention for any reason within 30 Days of scheduled procedure
14. Any percutaneous intervention, except for balloon valvuloplasty (BAV) within 1 month prior to implant procedure
15. Untreated clinically significant coronary artery disease requiring revascularization within 30 days before or after the study procedure
16. Acute myocardial infarction within 1 month prior to implant procedure
17. Previous TIA or stroke within 6 months prior to implant procedure
18. Active gastrointestinal (GI) bleeding within 3 months prior to implant procedure
19. Scheduled surgical or percutaneous procedure to be performed prior to 30 day visit
20. History of bleeding diathesis, coagulopathy, refusal of blood transfusions or severe anemia (Hb<8 g/dL)
21. Systolic pressure <80mmHg, cardiogenic shock, need for inotropic support or IABP
22. Primary hypertrophic obstructive cardiomyopathy (HOCM)
23. Active infection or endocarditis
24. Hepatic failure (> Child B)
25. Chronic renal dysfunction with serum creatinine > 3.0 mg/dL or renal dialysis
26. Neurological disease severely affecting ambulation, daily functioning, or dementia
27. Life expectancy < 12 months due to non-cardiac co-morbid conditions
28. Intolerance to aspirin, clopidogrel, contrast media, or porcine tissue and allergy to nickel
29. Pregnant or breast-feeding women
30. For other severe illnesses of the patient (e.g. active carcinoma), the investigator shall decide on an individual basis whether the patient is not to be included in the study
31. Currently participating in an investigational drug or another device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2017-04-17 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Primary Safety: freedom from all-cause mortality | 6 months post procedure
  freedom from all-cause mortality
Primary Device Performance:Procedure success in absence of MACCE | 30 days post procedure
  Procedure success in absence of MACCE

SECONDARY OUTCOMES:
Rate of clinical endpoints according to the Valve Academic Research Consortium (VARC 2) guidelines | 30 Days and month 12
  VARC 2 guidelines include different safety and efficacy endpoints like mortality, MI, stroke, etc.
Incidence of all cause mortality at 30 Days and 12 Months | 30 days and 12 months
  Incidence of all cause mortality at 30 Days and 12 Months
Freedom from MACCE at 30 Days, 6 Months and 12 Months | 30 Days, 6 Months and 12 Months
  Freedom from MACCE at 30 Days, 6 Months and 12 Months
Number of patients who have a Procedural success defined by a combination of criteria | procedure
  Procedural success defined as ACURATE neo™ at intended location with
Rate of device success | 7 days/ Discharge, 30 Days, 6 Months and at 12 Months
  Rate of device success
NYHA Functional Classification improvement | 30 Days, 6 Month and at 12 Months
  NYHA Functional Classification improvement
Echocardiographic assessment of valve performance (at 7 Days or Discharge, 30 Days, 6 Months, 12 Months) using a combination of measures | 7 Days or Discharge, 30 Days, 6 Months, 12 Months
  Echocardiographic assessment of valve performance (at 7 Days or Discharge, 30 Days, 6 Months, 12 Months) using a combination of measures

CONTACTS AND LOCATIONS:
Overall Officials: Markus Pr Schönburg, Prof.Dr.Med, Principal Investigator — Abteilung Herzchirurgie Kerckhoff-Klinik
Locations (7):
- Germany (7):
  - Kerckhoff-Klinik, Bad Nauheim
  - Krankenhausbetriebsgesellschaft, Bad Oeynhausen
  - Deutsched Herzzentrum Berlin, Berlin
  - Martin Luther University Halle Winttenberg, Halle
  - Universitätklinikum Hamburg Eppendorf, Hamburg
  - Herzentrum Leipzig GmbH, Leipzig
  - University Hospital Regensburg, Regensburg

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-requests.html).

REFERENCES:
- [Derived] Conradi L, Hilker M, Kempfert J, Borgermann J, Treede H, Holzhey DM, Schrofel H, Kim WK, Schaefer U, Walther T. Prospective multicentre evaluation of a novel, low-profile transapical delivery system for self-expandable transcatheter aortic valve implantation: 6-month outcomes. Eur J Cardiothorac Surg. 2018 Oct 1;54(4):762-767. doi: 10.1093/ejcts/ezy097. PMID 29554265